CLINICAL TRIAL: NCT01093560
Title: Fat Effects in Women With Metabolic Syndrome
Acronym: FEMMES II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Pathmaja Paramsothy, MD, MS, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 36899-D
Record Dates: First submitted 2010-03-18; First posted 2010-03-26 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; premenopausal women; fat feeding
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- young women with MetS (Experimental): 1. Saturated fat (control)
  2. n-3 Polyunsaturated fat (experimental)
  3. monounsaturated fat
  Interventions: Dietary Supplement: fat feeding

INTERVENTIONS:
Dietary Supplement: fat feeding — Each feeding will consist of 473 mL of nonfat milk and 50 gms oil. The oil will be high in saturated fat, monounsaturated fat or polyunsaturated fat.

SUMMARY:
Among 10 premenopausal women with Metabolic Syndrome:

Specific Aim 1: Compare the effects of acute fat feeding on flow mediated dilation (FMD) as measured by brachial artery reactivity among three fat challenges (saturated fat vs. monounsaturated fat (MUFA) vs. polyunsaturated fat (PUFA)at 4 hours post feeding. Hypothesis Saturated fat feeding will impair FMD but MUFA and PUFA feeding will not.

Specific Aim 2: Compare the effects of acute feeding on vascular inflammation as measured by VCAM and sICAM among three fat challenges at 3 1/2 hours post feeding.

Hypothesis: Saturated fat feeding will increase vascular inflammation but MUFA and PUFA will not.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* 18-50 years of age,
* Pre-menopausal,
* Weight stable for at least 3 months,
* Not planning to lose or gain weight for 3 months,
* Meets the following 3/5 criteria for metabolic syndrome:

  * increased blood sugar
  * increased blood fats (triglycerides),
  * increased blood pressure,
  * decreased good cholesterol (HDL-C).
  * increased waist circumference,

Exclusion Criteria:

* History of diabetes mellitus
* Fasting glucose ≥ 126 mg/dL
* History of cardiovascular disease (peripheral vascular disease, coronary artery disease, cerebrovascular disease)
* Pregnant or planning a pregnancy within the study period
* Fasting triglycerides > 500 mg/dL
* Currently taking lipid lowering medications**
* Oral or patch hormone contraception**
* Currently taking vaso-active (blood pressure) medications**
* SBP ≥ 140 and/or DBP ≥90 mm Hg or taking blood pressure lowering Rx
* Chronic use of aspirin (prn use is allowed)
* Chronic use of non-steroidal anti-inflammatory medications (prn use is allowed)
* Tobacco use within 6 months of starting study
* Participation in another clinical trial within the last 30 days
* History of active gall bladder disease
* History of digestive or malabsorptive disease requiring treatment or surgery
* Moderate to severe lactose intolerance
* Milk Allergy
* Walnut Allergy or Nut Allergy
* Coconut allergy

(**) Drugs within the following classifications are exclusionary: Lipid lowering, beta blockers, ACE inhibitors, angiotensin receptor blockers, diuretics, calcium channel blockers, alpha blockers, nitrates, hormone contraception includes patch or oral hormone contraception (Hormone containing IUDs or vaginal rings are okay)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilation at 4 hours post feeding | four hours
  4 hours

SECONDARY OUTCOMES:
Adhesion molecules (VCAM and sICAM) | 3 1/2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pathmaja Paramsothy, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States